CLINICAL TRIAL: NCT04949204
Title: Contextuele Analyse, Fysiologische Metingen en Machinaal Leren Voor Migraine en Clusterhoofdpijn (COPIMAC Studie)
Brief Title: Context-awareness, Physiological Monitoring, and Machine Learning in Migraine and Cluster Headache
Acronym: COPIMAC
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-07403
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Migraine; Cluster Headache
MeSH Terms: conditions — Migraine Disorders; Cluster Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migraine patients: Wearable wrist sensor + headache application on smartphone
  Interventions: Procedure: Wearable sensor detection
- Cluster Headache Patients: Wearable wrist sensor + headache application on smartphone
  Interventions: Procedure: Wearable sensor detection

INTERVENTIONS:
Procedure: Wearable sensor detection — Empatica E4 wearable wrist sensor

SUMMARY:
This is an observational, longitudinal cohort pilot study measuring physiological signals through wearable sensors combined with machine learning algorithms to detect behaviour, stress and headaches in patients with migraine and cluster headache.

DETAILED DESCRIPTION:
Migraine and cluster headache are among the most disabling headache conditions in humans. Both conditions have different phases such as the prodromal/premonitory phase, the aura phase, the headache phase and the postdromal phase. This pilot study examines the potential of wearable sensors combined with machine learning algorithms to investigate the biological changes over time in both conditions. Behaviour such as movement, sleep and activity will be monitored. Stress levels will be estimated through the wearable data combined with input from the patients. Participants will use a wearable device around the wrist and self-developed headache application for 21 days.

ELIGIBILITY:
Inclusion Criteria:

* migraine or cluster headache diagnosis based on ICHD 3 criteria
* at least 2 attacks each month
* onset of headache syndrome before the age of 50
* if multiple headache syndromes coexist: attacks are clearly distinguishable
* participant has smartphone that he/she wants to apply for this research

Exclusion Criteria:

* chronic migraine patients
* history of alcohol or illicit drug abuse
* significant medical comorbidity deemed by the investigator to interfere with the study
* use of betablockers
* participating in other academic or commercial trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Migraine or cluster headache patients
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Galvanic Skin Response changes | 21 days
  Changes in GSR through the different phases of the headache attacks

SECONDARY OUTCOMES:
Activity ratio | 21 days
  Activity ratio measurement through accelerometer data
Skin temperature | 21 days
  Skin temperature measurement through builtin thermometer

OTHER OUTCOMES:
Prevalence of premonitory symptoms | 21 days
Prevalence of cranial autonomic symptoms | 21 days
Prevalence of postdromal symptoms | 21 days
MSQv2.1 questionnaire | 21 days
  In migraine patients
MIDAS questionnaire | 21 days
  In migraine patients
SF20 | 21 days
  In migraine and cluster headache patients

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Ghent: Department of Neurology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vandenbussche N, Van Der Donckt J, De Brouwer M, Steenwinckel B, Stojchevska M, Ongenae F, Van Hoecke S, Paemeleire K. Patients with chronic cluster headache may show reduced activity energy expenditure on ambulatory wrist actigraphy recordings during daytime attacks. Brain Behav. 2024 Jan;14(1):e3360. doi: 10.1002/brb3.3360. PMID 38376015
- [Derived] De Brouwer M, Vandenbussche N, Steenwinckel B, Stojchevska M, Van Der Donckt J, Degraeve V, Vaneessen J, De Turck F, Volckaert B, Boon P, Paemeleire K, Van Hoecke S, Ongenae F. mBrain: towards the continuous follow-up and headache classification of primary headache disorder patients. BMC Med Inform Decis Mak. 2022 Mar 31;22(1):87. doi: 10.1186/s12911-022-01813-w. PMID 35361224